CLINICAL TRIAL: NCT00040287
Title: Theory-Based Interventions for Smoking and Obesity (Challenge) Trial
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: National Institute of Neurological Disorders and Stroke (NINDS) (NIH)
Allocation: Randomized | Purpose: Treatment
Other Study IDs: R01NS038441 (NIH)
Record Dates: First submitted 2002-06-24; First posted 2002-06-25 (Estimated); Last update posted 2007-05-17 (Estimated); Status verified 2007-05

CONDITIONS: Smoking; Obesity
Keywords: smoking; obesity; weight loss; smoking cessation; weight control
MeSH Terms: conditions — Smoking; Obesity; Weight Loss; Smoking Cessation

INTERVENTIONS:
Behavioral: smoking cessation program
Behavioral: weight control program

SUMMARY:
The purpose of this study is to examine a new theory for understanding the processes that govern behavior change by observing how people's beliefs and feelings about smoking cessation or weight loss change as they participate in smoking cessation or weight control programs. This study also seeks to improve the ability of treatment programs to help people maintain changes in their behavior.

DETAILED DESCRIPTION:
The goal of this clinical trial is to examine a new theory for understanding the processes that govern short-term versus long-term behavior change. The study will examine how people's beliefs and feelings about smoking cessation or weight loss change as they participate in either a smoking cessation program or a weight control program. Also, the study will improve the ability of treatment programs to help people maintain changes in their behavior. The project involves a series of two parallel investigations.

Study 1 tests the hypothesis that intervention methods that influence cost/benefit expectations related to quitting smoking and losing weight will have different effects on long-term smoking cessation and weight loss. The participants are randomly selected to treatment programs that induce heightened or realistic outcome expectations.

Study 2 tests the hypothesis that intervention methods that influence perceived satisfaction with behavior change will have different effects on long-term smoking cessation and weight loss. The participants are randomly selected to treatment programs that induce them to evaluate the consequences of behavior change either in comparison to past or ideal outcomes.

All of the intervention programs used in these studies are based on highly effective treatment procedures. The programs differ in how information about weight loss and smoking cessation is presented, how the participants are encouraged to think about their achievements during the treatment programs, and how much help is given to the participants in organizing their thoughts during the programs.

ELIGIBILITY:
Eligibility criteria for the smoking cessation studies were: between 18 and 60 years old, a minimum 2-year history of smoking, a current level of smoking > 10 cigarettes per day, and agreement to participate in the study.

Eligibility requirements for the weight loss studies were: between 18 and 60 years old, body mass index (weight/height2) > 27.0, 20 percent or more above desirable weight according to medical standards, and consent to participate.

Smokers and overweight persons were excluded if currently being treated by a physician for a serious physical or psychological disorder (e.g., heart disease, cancer, depression). Women were excluded if currently pregnant, pregnant in the last 6 months, or intending to become pregnant in the next 18 months. People who were overweight and who also smoked were considered eligible for participation in either weight loss or smoking cessation programs. However, they received treatment only for the particular behavior problem targeted by the study they chose to participate in.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1778
Dates: Start 1999-01

CONTACTS AND LOCATIONS:
Overall Officials: Robert Jeffery, Ph.D., Principal Investigator — University of Minnesota, Division of Epidemiology, School of Public Health
Locations (1):
- University of Minnesota, Division of Epidemiology, School of Public Health, Epidemiology Clinic Research Center, Suite 201, 1100 Washington Avenue South, Minneapolis, Minnesota, United States